CLINICAL TRIAL: NCT04128345
Title: Novel Multimodality Imaging Techniques for Neurosurgical Planning and Stereotactic Navigation in Lateral Skull Base Surgery: a Feasibility Study
Brief Title: Novel Multimodality Imaging for Navigation in Skull Base Surgery
Acronym: SBN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0661
Record Dates: First submitted 2019-09-18; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SBN arm: We will evaluate the feasibility of using an integrated navigation system incorporating pre-operative MRI and intraoperative ultrasound images
  Interventions: Device: Use of navigation system

INTERVENTIONS:
Device: Use of navigation system — Feasibility assessment of using an integrated navigation system incorporating advanced diffusion MRI, volumentric tumour representation and intraoperative ultrasound

SUMMARY:
Successful neurosurgery to remove tumours around the base of the skull, such as a vestibular schwannoma, depends on achieving maximal tumour removal whilst preserving crucial neurological functions such as facial movement, and maintaining quality of life.

Current techniques to direct surgery are based on the surgeon's expertise and knowledge of the relevant anatomy, supplemented by the use of electrical recording and stimulation of the facial nerve. However, it is often very difficult to visualise the nerve during surgery and facial nerve paralysis remains a potentially devastating complication of surgery.

Advanced imaging methods may be used to visualise important neural connections in the brain and computer-assisted processing can generate tumour maps from MRI and ultrasound scans. This study aims to utilise these technologies to develop a 3D navigation system for skull base surgery.

This study aims to develop a system that will combine MRI and intraoperative ultrasound imaging to enhance the surgeon's view of the tumour, facial nerve and other surrounding critical structures during surgery. This information will be made available in the navigation system in the operating room so that operations are more precise resulting in better tumour removal rates and fewer complications.

The system will be assessed during the treatment of 20 patients with vestibular schwannoma at the National Hospital for Neurology and Neurosurgery. This feasibility study will validate the different parts of the new system and help us design a future research study to determine its effectiveness in improving patient care.

This project will result in safer and more effective neurosurgery, with potential consequent financial savings for the NHS and the UK, in addition to marked improvements in the quality of life of patients and reduced dependency upon others.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-85 years
* Patients with a vestibular schwannoma who are scheduled for surgery
* Patients willing and able to provide written informed consent

Exclusion Criteria:

* Patients aged under 18 years of age or older than 85 years
* Previous, treated posterior fossa brain tumour(s)
* Previous ear or facial surgery on ipsilateral side of tumour
* Neurofibromatosis Type II
* Participation in other clinical trials
* Any contraindication for MR imaging
* Any contraindication for MR contrast agent administration
* Any contraindication for CT imaging
* Pregnancy or breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 - 85 years with a vestibular schwannoma who are scheduled for surgery and able to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
To assess the functionality and performance of a 3D surgical technical platform for integrating data from 3 different data sources (MRI, US and Neuronavigation data) in a clinical setting using a composite of quantitative and qualitative measurements | Data will be collected on the date of patients' routine surgical procedure, assessed on 1 day from the start time (hh:hh) of set-up of the 3d surgical platform to the end time (hh:hh) of surgery
  Composite of quantitative and qualitative measurements to assess the system's functionality and technical performance

SECONDARY OUTCOMES:
Correlation of electromyographic stimulation of facial nerve with preoperatively acquired diffusion imaging | A minimum of 9 time points (selected at random) during each surgical procedure, assessed on 1 day from the start time (hh:hh) to the end time (hh:hh) of surgery
  Stimulation response (binary outcome) and amplitude (mA)
Postoperative tumour volume on contrast-enhanced MRI and its correlation with the final intraoperative ultrasound measurement | Final intraoperative US volume vs post op MRI volume (within 3 months)
  Tumour volume (cm3) on MRI and US
Average duration of surgical procedure using 3D navigation system | From start time to end time of each surgical procedure, assessed on 1 day
  Time (hours)
Documentation of technical system issues and implemented solutions | From start time to end time of each surgical procedure, assessed on 1 day
  Documentation of technical system issues and implemented solutions (using qualitative research methods)

CONTACTS AND LOCATIONS:
Locations (1):
- University College London/University College London Hospitals Joint Research Office, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No